CLINICAL TRIAL: NCT07346651
Title: The Effect of Percussive Massage Therapy Using a Heat Therapy Attachment on Pain and Disability in Patients With Chronic Low Back Pain
Brief Title: Percussive Massage Therapy Using Heat Attachment in Chronic Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Arzu Razak Ozdinçler, Professor Doctor, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 39.2025fbu; 1919B012439024 (Other Grant/Funding Number: The Scientific and Technological Research Council of Türkiye (TÜBİTAK))
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Chronic Low Back Pain (CLBP)
Keywords: low back pain; percussive massage therapy; vibration; exercise
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Exercise; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This trial is assessor-blinded. The intervention will be delivered by study personnel who are not involved in outcome assessments. Outcome assessors will be unaware of group allocation. Participants will be instructed not to disclose their assigned group or any treatment details to the outcome assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percussive Massage Therapy (PMT) Group (Experimental): Participants assigned to the PMT group will receive conventional rehabilitation (exercise training + TENS) plus PMT. PMT will be administered after each conventional rehabilitation session, applied directly over the paravertebral muscles. Treatment will be delivered 5 days per week for 2 weeks, with 4 minutes applied to each side (8 minutes in total).
  Interventions: Device: Percussive Massage Therapy; Behavioral: Exercise Training (Conventional Rehabilitation); Device: Transcutaneous Electrical Nerve Stimulation (Conventional Rehabilitation)
- Control Group (Active Comparator): Participants assigned to the control group will receive a conventional rehabilitation program consisting of a supervised exercise program and Transcutaneous Electrical Nerve Stimulation (TENS). Treatment will be delivered 5 days per week for 2 weeks.
  Interventions: Behavioral: Exercise Training (Conventional Rehabilitation); Device: Transcutaneous Electrical Nerve Stimulation (Conventional Rehabilitation)

INTERVENTIONS:
Device: Percussive Massage Therapy — PMT will be delivered using a percussive massage therapy device (Therabody™, California, ABD) set to 1900 percussion per minute (31.67 Hz) with a heat-therapy attachment (50-55 °C), infrared LED light therapy enabled, and a 16-mm depth setting. Participants will be positioned prone with arms alongside the body. Following the conventional rehabilitation session, the thoracolumbar region will be exposed, and PMT will be applied in direct contact with the soft tissue over the paravertebral muscles, progressing from caudal to cranial. The therapist will move the device at a constant speed along a straight line to target the thoracolumbar fascia, performing repeated caudal-to-cranial and cranial-to-caudal passes (approximately 20 seconds per cycle) while maintaining consistent pressure using only the weight of the device. PMT will be applied for 8 minutes per session (4 minutes per side), 5 days per week for 2 weeks.
  Arms: Percussive Massage Therapy (PMT) Group
Behavioral: Exercise Training (Conventional Rehabilitation) — All participants will recieve a supervised exercise program including core stabilization and mobility/stretching exercises, delivered 5 days per week for 2 weeks (10 sessions). Exercise training will be delivered using brochures that include illustrations and written instructions to facilitate participants' learning of the exercises. The program includes eight exercises, each performed as 1 set of 10 repetitions, with appropriate interval between exercises. Exercises include supine abdominal drawing in maneuver, straight leg raise, bridge, upper and lower abdominal exercises (abdominal curl and heel slides), clamshell, cat-cow (also known as cat-camel), and child's pose.
Device: Transcutaneous Electrical Nerve Stimulation (Conventional Rehabilitation) — Burst TENS will be delivered using the Chattanooga® Intelect Advanced Stimulation Unit (Chattanooga, Tennessee, USA). It will be applied to the lumbar region. Four self-adhesive electrodes (50 mm × 50 mm) will be placed bilaterally, approximately 1.5 cm lateral to the spinous processes, in a symmetrical arrangement. Stimulation parameters will be 100 Hz pulse frequency, 2 Hz burst frequency, and 50-80 μs pulse duration. Current intensity will be set according to participant tolerance at a sensory level below the pain threshold. Each session will last 20 minutes.

SUMMARY:
Low back pain is a global problem that currently affects many people's participation in daily activities, and its prevalence has been increasing over the years. Exercise is among the most effective treatment approaches for reducing and preventing pain and disability related to low back pain. To enhance the effects of exercise, various adjunctive methods may be needed. Local vibration applications delivered through mechanical devices are offer practical and time-efficient application, which may reduce the physiotherapist's manual workload, while also providing potential benefits for patients with musculoskeletal pain. Therefore, the aim of this study is to investigate the effects of Percussive Massage Therapy (PMT) applied using a heat-therapy attachment on pain, disability, spinal mobility, health-related quality of life, kinesiophobia, and patient satisfaction in individuals with chronic low back pain.

Patients with chronic low back pain who meet the inclusion criteria will be randomly assigned to either the PMT group or the Control group (CG). All participants will receive a conventional rehabilitation program consisting of supervised exercise training and transcutaneous electrical nerve stimulation (TENS) for 2 weeks, 5 days per week, for approximately 45 to 60 minutes per day. The CG will receive only this conventional rehabilitation program. In addition, participants in the PMT group will receive PMT immediately after each conventional rehabilitation session, consisting of an 8-minute application (4 minutes per side) over the paravertebral muscles using a percussive massage therapy device.

Outcome measures will be assessed at baseline and post-treatment (end of week 2). Pain intensity will be evaluated using the Visual Analog Scale (VAS); disability using the Oswestry Disability Index (ODI); spinal flexibility using the finger-to-floor distance test; health-related quality of life using the Short Form-36v2 (SF-36v2); and kinesiophobia using the Tampa Scale for Kinesiophobia (TSK). Treatment satisfaction will be assessed post-treatment using the Global Perceived Effect Scale (GPE), and all data will be recorded on a data collection form.

DETAILED DESCRIPTION:
In 2020, low back pain affected an estimated 619 million people worldwide, and this number is projected to reach 843 million by 2050, with a disproportionate burden among socioeconomically disadvantaged populations. To avoid harmful and ineffective treatments, evidence supporting the safety, effectiveness, and cost-efficiency of interventions should be integrated into routine care, and greater investment in clinical research is needed to reduce the gap between research and clinical practice.

Clinical practice guidelines indicate that exercise is a primary non-invasive approach for reducing pain and disability in chronic low back pain. Adjunct non-pharmacological methods such as electrotherapy and massage are often used to enhance treatment effects. Although the evidence for vibration therapy is still emerging and has focused mainly on whole-body vibration, local vibration remains a promising but under-studied option for individuals with low back pain.

Local vibration can be delivered using different modalities, one of which is percussive massage therapy (PMT). PMT is applied via a mechanical device that delivers low-frequency pressure pulses to the skin, transmitting vibration to the underlying myofascial tissues. It is widely used as a low-cost and accessible adjunct for pain management, injury prevention, and rehabilitation. Previous studies have reported that vibration-based massage interventions are safe and well tolerated, and PMT has shown beneficial effects in neck pain and in selected low back pain populations, although evidence remains limited.

Soft tissue massage may alleviate pain by increasing local blood flow and oxygenation and by modulating neurophysiological pathways, including stimulation of large-diameter afferent fibers that can reduce pain perception via gate control mechanisms. Similarly, localized vibration can increase tissue perfusion, oxygen saturation, and temperature. PMT, which delivers low-frequency, localized mechanical pulses to myofascial tissues, may further influence pain through activation of mechanoreceptors and central pain-modulating pathways. These effects provide a rationale for investigating the impact of PMT delivered with a heat-therapy attachment on pain and disability in individuals with chronic low back pain.

Studies investigating mechanisms related to the effects of PMT applied to the low back have examined its potential effects on posture-related parameters, trigger points, and thoracolumbar fascia (TLF) characteristics, including echo intensity and thickness. Proposed mechanisms include reductions in myofascial stiffness through mechanical loading and heat-related changes that may influence tissue viscoelasticity, as well as neurophysiological effects that could reduce fascial tension and improve tissue extensibility. Acute PMT has been reported to increase tissue temperature and reduce TLF echo intensity and perceived stiffness, while TLF thickness appears largely unchanged across short- to longer-term observations in both healthy individuals and pationts with low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 to 55 years.
* Diagnosis of chronic low back pain confirmed by a physician (pain localized to the lumbar region, above the inferior gluteal folds and below the costal margin) with a duration of ≥ 3 months.
* Baseline pain intensity of 30-80 mm on the Visual Analog Scale (3 cm ≤ VAS ≤ 8 cm).

Exclusion Criteria:

* History of, or planned, surgery involving the low back or abdominal region.
* Malignancy, vertebral fracture, or other serious spinal pathology.
* Spinal injection or intervention within the past 3 months (e.g., epidural injection, facet joint steroid injection, neuroplasty).
* Long-term use of analgesic or corticosteroid medications that may affect musculoskeletal symptoms.
* Diagnosis of radiculopathy or neuropathy (with or without spinal canal stenosis).
* Cognitive impairment that would preclude providing informed consent.
* Significant structural spinal deformity (e.g., spondylolisthesis, congenital spinal deformities).
* Progressive neurological disorder affecting the lower limbs/spine or inflammatory spinal disease (e.g., axial spondyloarthritis), or cardiovascular instability.
* Pregnancy.
* Medical conditions contraindicating exercise participation

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Visual Analag Scale | Baseline, post-intervention (approximately 2 weeks)
  Paint intensity will be assessed using 10 cm Visual Analog Scale, ranging from no pain (0) to worst pain" (10). Participants will mark their perceived pain level on the scale; higher scores indicate greater pain intensity.
Oswestry Disability Index | Baseline, post-intervention (approximately 2 weeks)
  Disability will be assessed using the Oswestry Disability Index, version 2.0. The ODI is a self-administered questionnaire consisting of 10 sections, each scored from 0 to 5, with higher scores indicating greater disability in activities of daily living. The total score is converted to a percentage using the formula (total score × 100 / 50), yielding a range from 0 to 100. Scores are interpreted as follows: 0-20 minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound or symptom exaggeration/aggravation.

SECONDARY OUTCOMES:
Short Form-36v2 | Baseline, post intervention (approximately 2 weeks)
  Health-related quality of life will be assessed using the Turkish version of the Short Form-36 version 2 (SF-36v2). The SF-36v2 evaluates eight domains: Physical Functioning, Social Functioning, Role Physical, Role Emotional, Mental Health, Bodily Pain, General Health, and Vitality/Energy. Domain scores are calculated according to standard scoring procedures, with higher scores indicating better quality of life.
Tampa Scale for Kinesiophobia | Baseline, post-intervention (approximately 2 weeks)
  Kinesiophobia will be assessed using the Tampa Scale for Kinesiophobia (TSK). TSK is a 17-item questionnaire rated on a 4-point Likert scale. Items 4, 8, 12, and 16 are reverse-scored. The total score ranges from 17 to 68 with higher scores indicating greater kinesiophobia.
Finger-to-Floor Distance Test | Baseline, post-intervention (approximately 2 weeks)
  Spinal mobility and flexibility will be assessed using the finger-to-floor distance test. Participants will stand and bend forward as far as possible while keeping the knees extended and attempting to reach the floor. The vertical distance between the tip of the third finger and the floor will be measured and recorded. Lower values indicate greater flexibility.
Global Perceived Effect Scale | Post-intervention (approximately 2 weeks)
  Patient satisfaction will be assessed using the Global Perceived Effect (GPE) scale. The GPE is rated from -5 to +5, where -5 indicates "much worse," 0 indicates "no change," and +5 indicates "completely recovered." Higher scores indicate greater perceived improvement and satisfaction with treatment.
Adverse Events | During the 2-week intervention period
  Adverse events will be recorded throughout the 2-week intervention period using standardized adverse event reporting forms. Events will be documented as treatment-related or unrelated, and serious adverse events and contraindications to the intervention will be captured when applicable.

CONTACTS AND LOCATIONS:
Locations (1):
- Göztepe Prof. Dr. Süleyman Yalçın City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No